CLINICAL TRIAL: NCT04411901
Title: The Role of Vitamin D3 in Pediatric Bronchiectasis Severity( CF Versus Non CF Bronchioectasis)
Brief Title: The Role of Vitamin D3 in Pediatric Bronchiectasis Severity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Heba Omara (Other)
Responsible Party: Sponsor-Investigator, Heba Omara, Principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Original study
Record Dates: First submitted 2020-05-22; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Cystic Fibrosis and Non CF Bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vitamin D 3 (Experimental): oral vitamin D3 drops and tablets
  Interventions: Drug: Cholecalciferol (vitaminD3)

INTERVENTIONS:
Drug: Cholecalciferol (vitaminD3) — Theraputic vitamin D3 for CF and non CF bronchiectasis children

SUMMARY:
Vitamin D3 therapy was effective in decreasing the frequency of pulmonary exacerbations and preserving lung functions , thereby improving the disease severity even more in non CF than CF bronchiectasis patients

DETAILED DESCRIPTION:
Objectives: To compare the effect of vitamin D3 on modifying the disease severity in CF and non CF bronchiectasis pediatric patients.

Patients and Methods: This was a randomized clinical trial evaluating the role of oral vitamin D3 supplementation for 6 months in forty patients with CF and non CF bronchiectasis under the age of 18 years with vitamin D deficiency or insufficiency . The primary outcome was to reach the sufficient Vitamin D level. The secondary outcome was to follow up the frequency of pulmonary exacerbations and lung function after vitamin D3 supplementation.

ELIGIBILITY:
Inclusion Criteria:

* ages less than 18 years .
* Patients with documented diagnosis of CF (by the presence of a twice positive sweat chloride test and or paired CFTR DNA genetic mutations).
* Patients with non CF bronchiectasis diagnosed clinically and radiologically ( sweat chloride test negative) with a high resolution CT-confirmed diagnosis and clinical history consistent with bronchiectasis .
* Vitamin D deficient or insufficient CF and non CF bronchiectasis patients

Exclusion Criteria: if they had

* sufficient Vitamin D level .
* chronic lung diseases other than CF and non CF bronchiectasis , liver or renal diseases.
* reported taking vitamin-D supplements or steroid therapy in the last 6 weeks.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
reach sufficient vitamin D level | 6 months
  vitamin D more than 30 ng/dl
decrease disease severity | 6 months
  decrease excerbations and increase lung function

CONTACTS AND LOCATIONS:
Locations (1):
- Children hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No